CLINICAL TRIAL: NCT02410213
Title: A Multi-center, Open-label, Single Arm Study to Characterize the Pharmacokinetics and Pharmacodynamics Profile of Intravenous Ferric Carboxymaltose in Pediatric Subjects 1-17 Years Old With Iron Deficiency Anemia (IDA)
Brief Title: A Study to Characterize the PK and PD Profile of IV FCM in Pediatric Subjects 1-17 Years Old With IDA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT13036
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Iron Deficiency Anemia (IDA)
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: Eligible subjects were enrolled sequentially in Cohort 1 (FCM at 7.5 mg/kg with a maximum single dose of 750 mg) and Cohort 2 (FCM at 15 mg/kg with a maximum single dose of 750 mg). Enrollment in Cohort 2 was initiated only after all subjects in Cohort 1 completed 4 weeks of therapy and a Data and Safety Monitoring Board (DSMB) approved continuation.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ferric Carboxymaltose (FCM) (Experimental): FCM at 7.5 mg/kg or 15 mg/kg to a maximum single dose of 750 mg iron, whichever is smaller
  Interventions: Drug: Ferric Carboxymaltose (FCM)

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM)
  Other Names: Injectafer

SUMMARY:
This is a Phase II, open-label, non-randomized, multi-center, single arm study to characterize the pharmacokinetic and pharmacodynamics (PK/PD) profile of Ferric Carboxymaltose dosing in pediatric subjects with IDA after receiving either a 7.5 mg/kg or 15 mg/kg dose of Ferric Carboxymaltose.

DETAILED DESCRIPTION:
This is a Phase II, open-label, non-randomized, multi-center, single arm study to characterize the pharmacokinetic and pharmacodynamics (PK/PD) profile of Ferric Carboxymaltose dosing in pediatric subjects with IDA after receiving either a 7.5 mg/kg or 15 mg/kg dose of Ferric Carboxymaltose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 1 to 17 years of age with assent to participation and his/her parent or guardian is willing and able to sign the informed consent approved by the Independent Review Board / Ethics Committee.
* Screening TSAT < 20%
* Screening Hemoglobin < 11 g/dL
* For subjects who are receiving an erythropoietin stimulating agent (ESA): stable ESA therapy (+/- 20% of current dose) for > 8 weeks prior to the qualifying screening visit and no ESA dosing or product changes anticipated for the length of the trial

Exclusion Criteria:

* Known hypersensitivity reaction to any component of Ferric Carboxymaltose.
* Subject previously randomized and treated in this study or any other clinical study of Ferric Carboxymaltose (FCM or VIT-45).
* Body mass index (BMI) ≤ 5th percentile for age (see APPENDIX 2)
* Male or Female subject 1 year of age weighing < 12kg.
* History of acquired iron overload, hemochromatosis or other iron accumulation disorders.
* Chronic kidney disease subjects on hemodialysis.
* Screening Ferritin level > 300ng/mL
* Subjects with significant severe diseases of the liver, hemopoietic system, cardiovascular system, psychiatric disorder or other conditions which on the opinion of the investigator may place a subject at added risk.
* Any active infection.
* Known positive hepatitis B antigen (HBsAg) or hepatitis C viral antibody (HCV) with evidence of active hepatitis.
* Known positive HIV-1/HIV-2 antibodies (anti-HIV).
* Anemia due to reasons other than iron deficiency (i.e. hemoglobinopathy). Subjects treated with vitamin B12 or folic acid deficiency are permitted.
* Intravenous iron and /or blood transfusion in the 4 weeks prior to screening.
* Immunosuppressive therapy that may lead to anemia (i.e. cyclophosphamide, azathioprine, mycophenolate mofetil). Note steroid therapy is permitted.
* Administration and / or use of an investigational product (drug or device) within 30 days of screening.
* Alcohol or drug abuse within the past six months.
* Female subjects who are pregnant or lactating, or sexually active female who are of childbearing potential not willing to use an acceptable form of contraceptive precautions during the study.
* Subject is unable to comply with study assessments.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2017-01-22 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Poland (8):
  - Szpital Uniwersytecki Katedra i Klinika Pediatrii, Hematologii i Onkologii, Bydgoszcz
  - Zespół Opieki Zdrowotnej w Dębicy z siedzibą w Dębicy , Oddział Dziecięcy, Dębica
  - Uniwersytecki Szpital Dziecięcy w Krakowie, Oddział Pediatrii i Gastroenterologii (V), Krakow
  - Klinika Hematologii, Onkologii i Transplantologii Dziecięcej Uniwersytecki Szpital Dziecięcy w Lublinie, Lublin
  - Oddział Ogólnopediatryczny; Uniwersytecki Szpital Dziecięcy w Lublinie, Lublin
  - Indywidualna Specjalistyczna Praktyka lekarska z siedzibą w Rzeszowie, Rzeszów
  - Klinika Pediatrii, Hematologii i Onkologii Dziecięcej, Szczecin
  - Klinika Gastroenterologii, Hepatologii, Zaburzeń Odżywiania i Pediatrii, Warsaw
- Russia (2):
  - State Budgetary Educational Institution of Higher Professional Education "Ryazan State Medical University named after academician I.P. Pavlov" of the Ministry of Health of the Russian Federation, Ryazan
  - State Educational Institution of Higher Professional Education Saint Petersburg State Pediatric Medical Acamy of Ministry of Health and Social Development of the Russian Federation, Saint Petersburg

REFERENCES:
- [Derived] Korczowski B, Farrell C, Falone M, Blackman N, Rodgers T. Safety, pharmacokinetics, and pharmacodynamics of intravenous ferric carboxymaltose in children with iron deficiency anemia. Pediatr Res. 2023 Oct;94(4):1547-1554. doi: 10.1038/s41390-023-02644-9. Epub 2023 May 19. PMID 37208431

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Ferric Carboxymaltose (FCM) 7.5 mg/kg: FCM at 7.5 mg/kg to a maximum single dose of 750 mg iron, whichever is smaller
  Ferric Carboxymaltose (FCM)
- Cohort 2: Ferric Carboxymaltose (FCM) 15 mg/kg: FCM at 15mg/kg to a maximum single dose of 750mg iron, whichever is smaller
Period: Overall Study
Arm/Group | Cohort 1: Ferric Carboxymaltose (FCM) 7.5 mg/kg | Cohort 2: Ferric Carboxymaltose (FCM) 15 mg/kg
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ferric Carboxymaltose (FCM): FCM at 7.5 mg/kg or 15 mg/kg to a maximum single dose of 750 mg iron, whichever is smaller
  Ferric Carboxymaltose (FCM)
Arm/Group | Ferric Carboxymaltose (FCM)
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Eligible subjects were enrolled sequentially in Cohort 1 or Cohort 2, for a total of 35 subjects.
  years
    Cohort 1 (FCM at 7.5 mg/kg to a maximum of 750mg): number analyzed (Participants) | 16
    Cohort 1 (FCM at 7.5 mg/kg to a maximum of 750mg) | 9.1 (6.13)
    Cohort 2 (FCM at 15 mg/kg to a maximum of 750mg): number analyzed (Participants) | 19
    Cohort 2 (FCM at 15 mg/kg to a maximum of 750mg) | 10.3 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Eligible subjects were enrolled sequentially in Cohort 1 or Cohort 2, for a total of 35 subjects.
  Participants
    Cohort 1 (FCM at 7.5 mg/kg to a maximum of 750mg): number analyzed (Participants) | 16
    Cohort 1 (FCM at 7.5 mg/kg to a maximum of 750mg): Female | 10
    Cohort 1 (FCM at 7.5 mg/kg to a maximum of 750mg): Male | 6
    Cohort 2 (FCM at 15 mg/kg to a maximum of 750mg: number analyzed (Participants) | 19
    Cohort 2 (FCM at 15 mg/kg to a maximum of 750mg: Female | 9
    Cohort 2 (FCM at 15 mg/kg to a maximum of 750mg: Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Poland | 30
  Russia | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: Maximum observed serum concentration; obtained directly from the serum concentration-time profile.
Time Frame: prior to dosing and 1, 2, 6, 12, 48 and 72 hours post dosing
Population: In Cohort 1, pharmacokinetic parameter values are excluded for one subject due to anomalous and consistently high concentrations, and for one subject due to missing concentration data at 1 and 2 hours post-dose.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Cohort 1: Ferric Carboxymaltose (FCM) 7.5 mg: FCM at 7.5 mg/kg to a maximum single dose of 750 mg iron, whichever is smaller
  Ferric Carboxymaltose (FCM)
- Cohort 2: Ferric Carboxymaltose (FCM) 15 mg/kg: FCM at 15 mg/kg to a maximum single dose of 750 mg iron, whichever is smaller
Arm/Group | Cohort 1: Ferric Carboxymaltose (FCM) 7.5 mg | Cohort 2: Ferric Carboxymaltose (FCM) 15 mg/kg
Number analyzed (Participants) | 14 | 19
µg/mL | 157 (33.8) | 310 (13.9)

ADVERSE EVENTS:
Time Frame: Initial treatment with study drug through completion of day 35 (28 days post-dose for subjects who early terminated from the study).
Groups:
- Cohort 2: Ferric Carboxymaltose (FCM) 15 mg/kg: FCM at 15 mg/kg to a maximum single dose of 750 mg iron, whichever is smaller
  Ferric Carboxymaltose (FCM)
Arm/Group | Cohort 1: Ferric Carboxymaltose (FCM) 7.5 mg/kg | Cohort 2: Ferric Carboxymaltose (FCM) 15 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/19
Other Adverse Events (participants affected / at risk) | 9/16 | 12/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Ferric Carboxymaltose (FCM) 7.5 mg/kg (N=16) | Cohort 2: Ferric Carboxymaltose (FCM) 15 mg/kg (N=19)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Ferric Carboxymaltose (FCM) 7.5 mg/kg (N=16) | Cohort 2: Ferric Carboxymaltose (FCM) 15 mg/kg (N=19)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodentitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 2 (2)
Infusion site pruritus (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-10-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02410213/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02410213/SAP_001.pdf